CLINICAL TRIAL: NCT02115321
Title: A Phase II/III Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172 and MK-8742 in Subjects With Chronic Hepatitis C Virus Infection With Advanced Cirrhosis and Child-Pugh (CP)-B Hepatic Insufficiency
Brief Title: Study of Efficacy and Safety of Grazoprevir (MK-5172) + Elbasvir (MK-8742) in Chronic Hepatitis C Participants With Child-Pugh (CP)-B Hepatic Insufficiency (MK-5172-059)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-059; 2014-000672-25 (EudraCT Number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: CP-B GZR 50 mg + EBR 50 mg (Experimental): CP-B participants take GZR 50 mg + EBR 50 mg once daily (q.d.) by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- Part A: NC GZR 100 mg + EBR 50 mg (Experimental): NC participants take GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: MK-5172A
- Part B: CP-B GZR 100 mg + EBR 50 mg (Experimental): CP-B participants take GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: MK-5172A
- Part C: CP-B GZR 50 mg or 100 mg + EBR 50 mg (Experimental): CP-B participants take GZR 50 mg or GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks (GZR dose chosen based on results of Part A CP-B arm).
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: MK-5172A

INTERVENTIONS:
Drug: Grazoprevir — GZR was supplied as two 25 mg tablets in the Part A CP-B arm, or as either one GZR 100 mg tablet or one fixed-dose combination (FDC) tablet containing GZR 100 mg + EBR 50 mg in a single tablet (MK-5172A) in the Part A NC arm. GZR was taken q.d. by mouth.
  Other Names: MK-5172
Drug: Elbasvir — EBR was supplied as 50 mg tablets and was taken q.d. by mouth.
  Other Names: MK-8742
Drug: MK-5172A — MK-5172A FDC tablet containing GZR 100 mg + EBR 50 mg taken q.d. by mouth.
  Arms: Part A: NC GZR 100 mg + EBR 50 mg; Part B: CP-B GZR 100 mg + EBR 50 mg; Part C: CP-B GZR 50 mg or 100 mg + EBR 50 mg

SUMMARY:
This study is being done to evaluate the efficacy and safety of the drug combination grazoprevir (GZR; MK-5172) + elbasvir (EBR; MK-8742) in participants with chronic hepatitis C virus (HCV) genotype (GT) 1, 4, or 6 infection and who have cirrhosis and Child-Pugh (CP) score 7-9 moderate hepatic insufficiency (CP-B). The primary hypothesis is that the percentage of HCV-infected participants with hepatic insufficiency (the CP-B population) achieving sustained viral response (SVR) 12 weeks after the end of all treatment (SVR12) will be greater than 60%. Additionally, ten non-cirrhotic (NC) HCV-infected GT1 participants will also be given GZR + EBR at the beginning of the study; this will be done for the purpose of collecting plasma pharmacokinetic (PK) data in HCV GT1-infected participants who do not have hepatic insufficiency.

DETAILED DESCRIPTION:
The study will be conducted sequentially in 3 Parts. Each participant will participate in only one Part.

Participants will be enrolled in either Part A, Part B, or Part C:

* Part A: CP-B participants will receive GZR 50 mg+ EBR 50 mg; NC participants will receive GZR 100 mg/EBR 50 mg.
* Part B: CP-B participants will receive GZR 100 mg + EBR 50 mg.
* Part C: CP-B participants will receive either GZR 50 mg or 100 mg + EBR 50 mg. Study progression from Part A to Part B and from Part B to Part C will be based upon a review of safety and efficacy in Parts A and B, respectively. Depending upon safety and efficacy in Part A, the study may progress directly from Part A to Part C using GZR 50 mg + EBR 50 mg, without performing Part B.

ELIGIBILITY:
Inclusion criteria:

* Has documented chronic HCV GT1 infection (for Arm 4 participants may have GT4 or GT6 infection) with no evidence of non-typable or mixed genotype infection
* Has clinical evidence of hepatic cirrhosis with a score on the Child-Pugh scale from 7 to 9 and not anticipated to receive a liver transplant within the next 36 weeks (for Arm 1, Arm 3, and Arm 4)
* Has no evidence of cirrhosis (only for Arm 2 )
* Agrees to remain truly abstinent or use (or have their partner use) an acceptable method of birth control from at least 2 weeks prior to Day 1 and continue until at least 14 days after last dose of study drug, or longer if dictated by local regulations

Exclusion criteria:

* Is co-infected with hepatitis B virus or human immunodeficiency virus (HIV)
* Has previously received direct-acting antiviral therapy for HCV
* Has a history of malignancy <=5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or under evaluation for other active or suspected malignancy
* Has cirrhosis and liver imaging results within 4 weeks prior to screening showing evidence of hepatocellular carcinoma (HCC), or is under evaluation for HCC
* Is currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study
* Has clinically-relevant drug or alcohol abuse within 12 months of screening
* Is pregnant or breast-feeding, or expecting to conceive or donate eggs or sperm from at least 2 weeks prior to Day 1 and continue throughout treatment and follow up, or longer if dictated by local regulations
* Has received organ transplants (including hematopoietic stem cell transplants) other than cornea and hair
* Has poor venous access
* Has a history of gastric surgery (e.g., stapling, bypass) or history of malabsorption disorders (e.g., celiac sprue disease)
* Requires, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
* Has evidence or history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2015-03-05 (Actual); Study Completion 2015-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Jacobson IM, Poordad F, Firpi-Morell R, Everson GT, Verna EC, Bhanja S, Hwang P, Caro L, Robertson M, Charles ED, Platt H. Elbasvir/Grazoprevir in People With Hepatitis C Genotype 1 Infection and Child-Pugh Class B Cirrhosis: The C-SALT Study. Clin Transl Gastroenterol. 2019 Apr;10(4):e00007. doi: 10.14309/ctg.0000000000000007. PMID 30939489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The screening period lasted for 60 days. Recruitment was halted after enrolling participants in the two Part A arms, as the current clinical development plan is focused on a fixed-dose combination (FDC) product containing grazoprevir (GZR) 100 mg and elbasvir (EBR) 50 mg. No participants were enrolled in Parts B or C.
Groups:
- Part A: CP-B GZR 50 mg + EBR 50 mg: Child-Pugh score 7 to 9 (CP-B) participants take GZR 50 mg + EBR 50 mg once daily (q.d.) by mouth for 12 weeks.
- Part A: NC GZR 100 mg + EBR 50 mg: Non-cirrhotic (NC) participants take GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks.
Period: Overall Study
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + EBR 50 mg
Started | 30 | 10
Completed | 29 | 10
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: CP-B GZR 50 mg + EBR 50 mg: CP-B participants take GZR 50 mg + EBR 50 mg q.d. by mouth for 12 weeks.
- Part A: NC GZR 100 mg + ER 50 mg: NC participants take GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (7.0) | 60.4 (5.3) | 58.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 17 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Viral Response 12 Weeks After Completing Study Therapy (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) levels below the lower limit of quantification (LLoQ) 12 weeks after completing study therapy. HCV RNA was measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay which has a LLoQ of 15 IU/mL and a limit of detection of 15 IU/mL.
Time Frame: Week 24
Population: The Full Analysis Set (FAS) consists of all randomized participants who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 30 | 10
Percentage of participants | 90.0 [73.5 to 97.9] | 100.0 [69.2 to 100.0]

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE) During Treatment and First 14 Follow-up Days
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 weeks
Population: The All Participants as Treated (APaT) population consisted of all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 30 | 10
Number of participants | 25 | 8

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 12 weeks
Population: The APaT population consisted of all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 30 | 10
Number of participants | 0 | 0

4. Secondary Outcome: Mean Change From Baseline in Model for End-Stage Liver Disease (MELD) Scores in CP-B Participants
Description: The MELD score provides an objective and granular assessment of liver improvement as a continuous variable. The calculation of MELD score is based on three biochemical variables (serum bilirubin, creatinine and international normalized ratio [INR] of prothrombin time). The MELD equation is as follows: 9.57 x ln(creatinine mg/dL) +3.78 x ln(bilirubin mg/dL) +11.2 x ln (INR) + 6.43. Scores are multiplied by 10 and rounded to the nearest whole number and range from 6 (less ill) to 40 (gravely ill). MELD scores were determined at Baseline (Day 1) and again at Week 12, Follow-up (FU) Week 12 (Week 24), and FU Week 24 (Week 36). Change from baseline in MELD score = Post-baseline MELD score - baseline MELD score.
Time Frame: Baseline and Weeks 12, 24, and 36
Population: All CP-B participants in the FAS (all randomized participants who received at least one dose of study medication) with available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 30 | 0
Units on a scale
  Week 12 (n=30) | -0.67 (1.35) |
  FU Week 12 (Week 24) [n=29] | -0.38 (1.74) |
  FU Week 24 (Week 36) [n=29] | -0.34 (3.15) |

5. Secondary Outcome: Percentage of Participants With HCV RNA Undetectable at Weeks 2, 4, and 12
Description: HCV RNA was measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay which has a LLoQ of 15 IU/mL and a limit of detection of 15 IU/mL.
Time Frame: Week 2, 4, and 12
Population: Per protocol, this measure was to be determined in Arm 4 (Part C); however, enrollment was halted after Part A and thus no data are available.
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With HCV RNA <LLoQ at Weeks 2, 4, and 12
Description: as for outcome 5
Time Frame: Weeks 2, 4, and 12
Population: as for outcome 5
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving Sustained Viral Response 4 Weeks After Completing Study Therapy (SVR4)
Description: SVR4 was defined as HCV RNA levels <LLoQ 4 weeks after completing study therapy. HCV RNA was measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay which has a LLoQ of 15 IU/mL and a limit of detection of 15 IU/mL.
Time Frame: Week 16
Population: The FAS consists of all randomized participants who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 30 | 10
Percentage of participants | 93.3 [77.9 to 99.2] | 100.0 [69.2 to 100.0]

8. Secondary Outcome: Percentage of Participants Achieving Sustained Viral Response 24 Weeks After Completing Study Therapy (SVR24)
Description: SVR24 was defined as HCV RNA levels <LLoQ 24 weeks after completing study therapy. HCV RNA was measured with the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay which has a LLoQ of 15 IU/mL and a limit of detection of 15 IU/mL.
Time Frame: Week 36
Population: The FAS consists of all randomized participants who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CP-B GZR 50 mg + EBR 50 mg | Part A: NC GZR 100 mg + ER 50 mg
Number analyzed (Participants) | 30 | 10
Percentage of participants | 90.0 [73.5 to 97.9] | 100.0 [69.2 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to 36 weeks.
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Groups:
- CP-B: GZR 50 mg + EBR 50 mg for 12 Weeks: CP-B participants take GZR 50 mg + EBR 50 mg q.d. by mouth for 12 weeks.
- Non-cirrhotic: GZR 100 mg + EBR 50 mg for 12 Weeks: NC participants take GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks.
Arm/Group | CP-B: GZR 50 mg + EBR 50 mg for 12 Weeks | Non-cirrhotic: GZR 100 mg + EBR 50 mg for 12 Weeks
Serious Adverse Events (participants affected / at risk) | 5/30 | 0/10
Other Adverse Events (participants affected / at risk) | 20/30 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CP-B: GZR 50 mg + EBR 50 mg for 12 Weeks (N=30) | Non-cirrhotic: GZR 100 mg + EBR 50 mg for 12 Weeks (N=10)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CP-B: GZR 50 mg + EBR 50 mg for 12 Weeks (N=30) | Non-cirrhotic: GZR 100 mg + EBR 50 mg for 12 Weeks (N=10)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 9 (11) | 3 (3)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (6)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.